CLINICAL TRIAL: NCT04140240
Title: Effect of Progressive Muscle Relaxation Training on Menopause Symptom Management and Quality of Life
Brief Title: Menopause Symptom Management in Perimenopause and Postmenopausal Period
Acronym: Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Gülşen Ak Sözer, lecturer, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Akd04050
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Menopause
Keywords: menopause management; progressive muscle relaxation; nursing

STUDY DESIGN:
Intervention Model Description: Parallel Assignment a experimental design with pre test and post test
Who Masked: Outcomes Assessor
Masking Description: Parallel Assignment a experimental design with pre test and post test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Experimental: İntervention group
  Interventions: Behavioral: intervention group
- Control group (No Intervention): Control group: No intervention

INTERVENTIONS:
Behavioral: intervention group — Parallel Assignment a experimental design with pre test and post test
  Arms: İntervention group

SUMMARY:
Aim:The aim of this study is to relieve menopause symptoms and improve quality of life by applying progressive muscle relaxation exercises to women in perimenopause and postmenopausal period.

Method: This study was planned as a pre-test, post-test, semi-interventional and control group study in order to relieve menopausal symptoms and to evaluate the effect on improving quality of life by applying progressive muscle relaxation exercises to women in perimenopause and postmenopausal period.

In the study, Individual Information Form, Menopause Symptom Rating Scale, Menopause Specific Quality of Life Scale were used to collect data.

The intervention group consisted of female students enrolled in GeroAtlas60 + Refresher University, which is a project of the Department of Gerontology, Faculty of Health Sciences, Akdeniz University. The Control group consisted of female students enrolled in the Mediterranean Family Health and Education Association. All female students who accepted to participate in the study and who met the inclusion criteria were included in the study. At the beginning of the study, pre-tests were applied to all participants. After 11 weeks of progressive muscle relaxation exercises, final tests were applied to the intervention group. The control group also underwent post-tests 11 weeks after any intervention. Progressive muscle relaxation exercises were then performed. After the researcher's explanation, the participants filled in the data collection forms themselves.

The post test data was collected in Jun 2019. The data will be entered in the SPSS file and the analysis of the data will be performed in the next stage.

DETAILED DESCRIPTION:
This study was conducted as a pre-test, post-test, semi-interventional and control group study to evaluate the effect of progressive muscle relaxation exercises on perimenopausal and postmenopausal women to relieve menopause symptoms and improve quality of life.

According to the World Health Organization, menopause is defined as a permanent termination of menstruation due to loss of ovarian activity . Menopause is a period of life from which the reproductive ability is lost, due to the decline in ovarian function of women. If menstruation is not observed for one year at the end of the reproductive period, menopause is considered to have started. Menopausal symptoms begin to appear in the premenopausal period and the effects continue in the postmenopausal period.

It is stated that symptoms seen in perimenopausal and post menopausal period adversely affect the quality of life of women. According to the results of the study, progressive relaxation exercises in perimenopause and postmenopausal women alleviate and relieve stress, anxiety and depression, pain, hot flash, and regulate blood pressure and pulse sleep.

Ethics committee approval and institutional permissions were obtained before starting the study. Written and verbal consent was obtained from all participants. In the study, Individual Information form, Menopause Symptom Rating Scale, Menopause Specific Quality of Life Scale were used to collect data. These data collection tools were used in the pre-test and post-test.

Women students who were registered to GeroAtlas60 + Refresher University of Akdeniz University Faculty of Health Sciences Department of Gerontology were appointed as an intervention group by lot method. Female students who accepted to participate in the study were divided into five groups and pre-tests were performed. The intervention group received 45 minutes of menopause symptom management training twice a week for two weeks. Then, 45 minutes of progressive muscle relaxation exercises were performed. In the first session, the participants were given a booklet of menopause management and progressive muscle relaxation exercises prepared by the researchers. At the end of the two-week learning process, the participants were given Progressive Muscle Relaxation Exercise Guide and Progressive Muscle Relaxation Exercise Calendar. At the same time, audio recording including Menopause Management and Progressive Muscle Relaxation Exercise application, which the researcher recorded by himself, was sent via wat's up. Reminder messages were sent to the participants via wta's up to remind them to come on the application days, the application to be held in the evening and do it themselves at home.Participants performed Progressive Muscle Relaxation Exercise two days a week in the presence of researchers. They recorded the voice of the researcher at home every other day. They marked their practice on the Progressive Muscle Relaxation Exercise Calendar for 11 weeks. This marked calendar was withdrawn from the participants at the end of the 11-week practice. After 11 weeks of progressive muscle relaxation exercises, post tests were applied to the intervention group. The control group also underwent post-tests 11 weeks after any intervention. Progressive muscle relaxation exercises were then performed. After the researcher's explanation, the participants filled in the data collection forms themselves.

The post test data was collected in Jun 2019. The data will be entered in the SPSS file and the analysis of the data will be performed in the next stage.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-65 years
* Not having menstruated during the last year
* To be at least primary school graduate
* To have a smart mobile phone
* Menopause symptom rating scale score of 15 and above

Exclusion Criteria:

* Being under 40,
* Being over 65 years of age,
* To use hormone replacement therapy for menopause symptoms in the last six months and during the study period,
* Use complementary therapy or progressive muscle relaxation exercises in the last two months for menopausal symptoms.
* No hearing impairment
* Being diagnosed with psychiatric illness

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale-MRS | 11 weeks
  Menopause Rating Scale, was first developed by Schneider et al. in 1992 to measure the severity of menopausal symptoms and their impact on quality of life. The Turkish validity and reliability of the scale was made by Gürkan (Gürkan, 2005). The total score of the scale is calculated based on the scores given for each item. The minimum score that can be obtained from the scale is 0 and the maximum score is 44. The increase in the total score obtained from the scale indicates the increase in the severity of the complaints on the one hand and the negative effect on the quality of life on the other. The 11-week progressive muscle relaxation exercises program was applied only to the intervention group. The statistically significant decrease in the mean scores of menopause rating scale in the post test in the intervention group is the success criterion of the study. Significance level is determined at p <0.05 in the analyzes.

SECONDARY OUTCOMES:
The Menopause Specific Quality of Life Questionnaire-MENQOL | 11 weeks
  Hilditch et al. (1996) to assess the quality of life of women in menopausal period and was standardized. Its validity and reliability in Turkish was made by Kharbouch and Şahin (2007). The Menopausal Quality of Life Scale is a Likert-type scale with 29 questions. As the score increases, the severity of the complaint increases. The lowest score that can be obtained from the total of the scale is 0 and the highest score (29X6) is 154.. However, the total score is not evaluated. MENQOL consists of four sub-scale. The higher the scores, the lower the quality of life. At the end of 11 weeks of progressive muscle relaxation exercise, scores are expected to decrease significantly in the intervention group. The significant decrease in post test scores as a result of the intervention is the success criteria of the study. Significance level is set at p<0.05 in analyzes.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Ege, professor, Study Director — Necmettin Erbakan University, Konya
Locations (1):
- Gülşen Ak Sözer, Antalya, Pınarbaşı Neighborhood, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Can Gürkan Ö; Menopoz Semptomlarını Değerlendirme Ölçeğinin Türkçe Formunun Güvenirlik ve Geçerliliği, Hemşirelik Forumu, sf:30-35, Mayıs-Haziran 2005.
- [Background] Kharbouch SB,Şahin Determination of the Quality of Life During Menopausal Stages. İ.Ü.F.N. Hem. Derg. 15 (59) : 82-90, 2007
- [Background] Chaudhuri A, Ray M, Saldanha D, Sarkar SK. Effects of progressive muscle relaxation on postmenopausal stress. Journal of the Scientifi c Society 42 (2): 62-67, 2015
- [Background] Kaur P, Kaur S, Shanmugam S, Kang M. Efficacy of Yoga versus Relaxation Techniques on Climacteric Symptoms of Perimenopausal women. IOSR Journal of Dental and Medical Sciences (IOSR-JDMS) 13( 7): 32-42, 2014. www.iosrjournals.org
- [Result] Johnson A, Roberts L, Elkins G. Complementary and Alternative Medicine for Menopause. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19829380. doi: 10.1177/2515690X19829380. PMID 30868921
- [Result] Schneider HP, Heinemann LA, Rosemeier HP, Potthoff P, Behre HM. The Menopause Rating Scale (MRS): reliability of scores of menopausal complaints. Climacteric. 2000 Mar;3(1):59-64. doi: 10.3109/13697130009167600. PMID 11910611
- [Result] Heinemann LA, Potthoff P, Schneider HP. International versions of the Menopause Rating Scale (MRS). Health Qual Life Outcomes. 2003 Jul 30;1:28. doi: 10.1186/1477-7525-1-28. PMID 12914663
- [Result] Tao M, Shao H, Li C, Teng Y. Correlation between the modified Kupperman Index and the Menopause Rating Scale in Chinese women. Patient Prefer Adherence. 2013;7:223-9. doi: 10.2147/PPA.S42852. Epub 2013 Mar 20. PMID 23569361
- [Result] Saensak S, Vutyavanich T, Somboonporn W, Srisurapanont M. Modified relaxation technique for treating hypertension in Thai postmenopausal women. J Multidiscip Healthc. 2013 Oct 3;6:373-8. doi: 10.2147/JMDH.S51580. eCollection 2013. PMID 24124377
- [Result] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630